CLINICAL TRIAL: NCT07247721
Title: Comparison of the Effects of Transcutaneous vs. Percutaneous Electrical Nerve Stimulation on the Sensorimotor System of the Radial Nerve in Healthy Volunteers
Brief Title: Transcutaneous vs Percutaneous Electrical Stimulation of the Radial Nerve
Acronym: TENS vs PENS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GIFTO-TENSvsPENS-2025
Record Dates: First submitted 2025-11-15; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pain Modulation; Sensorimotor Function; Nerve Stimulation
Keywords: Transcutaneous Electrical Nerve Stimulation; Percutaneous Electrical Nerve Stimulation; Low-Frequency Stimulation
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Transcutaneous Electrical Nerve Stimulation (TENS) (Active Comparator): Participants will receive one session of Transcutaneous Electrical Nerve Stimulation (TENS) applied over the radial nerve using surface electrodes. Stimulation parameters: 2 Hertz (Hz) frequency, 250 microseconds (µs) pulse width, and intensity set at the individual tolerance threshold for 20 minutes.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Percutaneous Electrical Nerve Stimulation (PENS) (Active Comparator): Participants will receive one session of Percutaneous Electrical Nerve Stimulation (PENS). A sterile 0.30 × 50 millimeter (mm) needle will be inserted near the radial nerve under ultrasound guidance. Stimulation parameters: 2 Hertz (Hz) frequency, 250 microseconds (µs) pulse width, and intensity set at the individual tolerance threshold for 20 minutes.
  Interventions: Device: Percutaneous Electrical Nerve Stimulation (PENS)
- Sham TENS (Sham Comparator): Participants will undergo a sham Transcutaneous Electrical Nerve Stimulation (TENS) procedure identical in setup and duration to the active TENS group. Electrodes will be placed in the same positions, and the current intensity will be increased for about 30 seconds until a strong but comfortable tingling is felt, then gradually reduced to 0 milliamperes (mA). The electrodes will remain in place for 20 minutes to mimic the active procedure. Neither participants nor evaluators will have visual access to the device display.
  Participants will also receive a placebo needle intervention, consisting of a non-penetrating sham needle applied to the same anatomical region without skin insertion. This procedure mimics the sensation of needling but does not break the skin or produce physiological effects.
  Interventions: Device: Sham Transcutaneous Electrical Nerve Stimulation
- Sham PENS (Sham Comparator): Participants will undergo a sham Percutaneous Electrical Nerve Stimulation (PENS) procedure. A real sterile acupuncture needle (0.30 × 50 millimeters (mm)) will be inserted at the same anatomical location used in the active PENS group, following the same ultrasound-guided procedure. The stimulator will remain switched off, following the same procedure used in the sham TENS group: the intensity will be increased for approximately 30 seconds until a comfortable tingling sensation is perceived and then gradually reduced to 0 milliamperes (mA), ensuring that no real stimulation is delivered.
  The needle will remain in place for 20 minutes to mimic the duration and setup of the active treatment.
  Interventions: Device: Sham Percutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Participants will receive one 20-minute session of Transcutaneous Electrical Nerve Stimulation (TENS) applied over the radial nerve of the non-dominant forearm. Two surface electrodes will be placed under ultrasound guidance (General Electric (GE) Logiq P9), longitudinally along the nerve path, approximately 5-8 centimeters (cm) proximal and distal to the lateral epicondyle. Stimulation parameters will consist of a biphasic symmetrical current at 2 Hertz (Hz) frequency, 250 microseconds (µs) pulse width, and an intensity adjusted to the maximum tolerable level without pain. The stimulator used will be an ENRAF NONIUS Endomed 484 (Madrid, Spain). Participants will remain in a supine position with the forearm supported in a prone posture. In addition, participants will receive a placebo needle intervention, consisting of a non-penetrating sham needle applied to the same anatomical region without skin insertion. This procedure mimics the sensation of needling but does not break the skin o
  Arms: Transcutaneous Electrical Nerve Stimulation (TENS)
Device: Percutaneous Electrical Nerve Stimulation (PENS) — Participants will receive one 20-minute session of Percutaneous Electrical Nerve Stimulation (PENS) targeting the radial nerve of the non-dominant forearm. A sterile 0.30 × 50 millimeter (mm) acupuncture needle will be inserted under ultrasound guidance (General Electric (GE) Logiq P9, General Electric Healthcare, Milwaukee, WI, USA) approximately 1-2 mm from the radial nerve, at a depth of 2-3 centimeters (cm), avoiding direct contact. A surface electrode will be placed 2.5 cm distal and 1 cm cranial to the needle. Stimulation parameters: biphasic current, 2 Hertz (Hz) frequency, 250 microseconds (µs) pulse width, and intensity adjusted to the maximum tolerable level without pain. The stimulator used will be an ENRAF NONIUS Endomed 484 (Madrid, Spain). Participants will remain in a supine position with the forearm supported in a prone posture.
  Arms: Percutaneous Electrical Nerve Stimulation (PENS)
Device: Sham Transcutaneous Electrical Nerve Stimulation — Participants will undergo a sham Transcutaneous Electrical Nerve Stimulation (TENS) procedure identical in setup and duration to the active TENS group. Two surface electrodes will be placed under ultrasound guidance (General Electric (GE) Logiq P9) along the nerve path, 5-8 cm proximal and distal, and the current will be increased for ~30 seconds until a strong but comfortable tingling is felt, then reduced to 0 milliamperes (mA). The electrodes will remain in place for 20 minutes to mimic the active procedure. The stimulator (ENRAF NONIUS Endomed 484) will remain on but deliver no current. Neither participants nor evaluators will have visual access to the device display to maintain blinding. Participants will also receive a placebo needle intervention, consisting of a non-penetrating sham needle applied to the same anatomical region without skin insertion. This procedure mimics the sensation of needling but does not break the skin or produce physiological effects.
  Arms: Sham TENS
Device: Sham Percutaneous Electrical Nerve Stimulation — Participants will undergo a sham Percutaneous Electrical Nerve Stimulation (PENS) procedure identical in setup and duration to the active PENS group. A sterile needle (0.30 × 50 millimeters (mm)) will be inserted under ultrasound guidance (General Electric (GE) Logiq P9, General Electric Healthcare, Milwaukee, WI, USA) at the same anatomical site and depth as in the active PENS group. However, no electrical current will be applied. The stimulator (ENRAF NONIUS Endomed 484) will remain on but disconnected from the needle to maintain participant blinding. Neither participants nor evaluators will have visual access to the device screen. Total session duration: 20 minutes.
  Arms: Sham PENS

SUMMARY:
This study aims to compare the effects of two types of electrical nerve stimulation techniques-Transcutaneous Electrical Nerve Stimulation (TENS) and Percutaneous Electrical Nerve Stimulation (PENS)-on the sensory and motor components of the radial nerve in healthy volunteers.

Transcutaneous Electrical Nerve Stimulation (TENS) is a non-invasive, low-cost, and widely used electrotherapy technique that applies electrical currents through surface electrodes on the skin to relieve pain. Percutaneous Electrical Nerve Stimulation (PENS) is a minimally invasive technique that delivers the electrical current through fine needles inserted near a peripheral nerve, potentially producing stronger physiological effects.

In this randomized, double-blind controlled clinical trial, 120 healthy participants aged 18-60 years will be randomly assigned to one of four groups:

Transcutaneous Electrical Nerve Stimulation (TENS)

Percutaneous Electrical Nerve Stimulation (PENS)

Sham Transcutaneous Electrical Nerve Stimulation (TENS) (placebo)

Sham Percutaneous Electrical Nerve Stimulation (placebo)

Each participant will receive one 20-minute stimulation session. Outcomes will include:

Pressure pain threshold (PPT) (measured with an algometer),

Thermal pain threshold (measured with a thermode),

Maximal Isometric wrist extensor strength (measured with a hand-held dynamometer).

The goal is to determine whether Percutaneous Electrical Nerve Stimulation (PENS) produces greater changes in sensory and motor parameters than Transcutaneous Electrical Nerve Stimulation (TENS) and to evaluate differences compared to placebo. This research will improve understanding of the physiological effects of these commonly used electrotherapy modalities and support evidence-based decision-making in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged between 18 and 60 years.
* No history of musculoskeletal or neurological disorders.
* No alterations in sensitivity in the upper limb.
* Not taking any medication in the previous two weeks.
* Able to understand the study procedures and provide informed consent.

Exclusion Criteria:

* Any neurological or neuromuscular disease.
* History of upper limb trauma, surgery, or persistent pain.
* Contraindications to electrical stimulation or invasive techniques.
* Presence of cardiac pacemaker, epilepsy, diabetes, cancer, or cardiovascular disease.
* Skin lesions or infections in the stimulation area.
* Pregnancy or suspected pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Threshold (PPT) | Baseline and immediately post-intervention
  Description: It will be assessed as an indirect measure of the effect on the Aδ sensory fibers of the radial nerve. To record the mechanical pain threshold, a point will be marked on the dorsal surface of the trapeziometacarpal joint. A digital algometer with an increment scale of 0.1 Newtons (N) (Wagner Instruments, model FDIX) and a circular probe of 1 centimeter (cm) in diameter will be used. Once the probe is placed perpendicular to the skin, pressure will be increased at a rate of approximately 5 Newtons per second (N/s). Three measurements will be taken, with 15-second intervals between them, and the mean of the three values will be recorded as the pressure pain threshold. The reproducibility and reliability of pressure algometry to measure pressure pain threshold have been demonstrated in previous studies.
Thermal Pain Threshold | Baseline and immediately post-intervention
  Thermal pain threshold will be assessed as an indirect measure of the effect on unmyelinated C-type sensory fibers of the radial nerve. Hot stimuli will be applied to the dorsal area of the second metacarpal (radial nerve dermatome) using a 9 square centimeters (cm²) Peltier thermode (TSA 2, MEDOC, Israel). Three ascending temperature ramps will be performed with one-minute intervals. The heat pain threshold will be determined by the method of limits, and the average of the three measurements will be recorded. Baseline temperature: 32 degrees Celsius (°C); increase rate: 1 degree Celsius per second (°C/s); decrease rate: 3 °C/s. Participants will press a button with the contralateral hand when the heat becomes painful, triggering automatic cooling. For safety, a 50 °C cutoff temperature will be used. Prior to testing, a familiarization trial will be conducted on the dominant hand over the first and second metacarpals.

SECONDARY OUTCOMES:
Maximal Isometric Wrist Extensor Strength | Baseline and immediately post-intervention
  It will be assessed as an indirect measure of the blockade of motor fibers (Aα motoneurons) of the radial nerve. Maximal isometric wrist extensor strength will be measured using a hand-held dynamometer (MicroFET 2, Hoggan Scientific, USA) following Méndez-Rebolledo et al. protocol. Subject position: supine, shoulder at 0° abduction, elbow at 0° flexion, forearm fully pronated, and wrist at 30° flexion with fingers extended. Evaluator position: standing, thighs touching the table; upper hand stabilizes the forearm above the styloid processes, lower hand holds the dynamometer over the distal third of the metacarpals. Stabilization: provided by the upper hand. Adapter: large flat type. Dynamometer placement: over metacarpal heads. Execution: three maximal isometric contractions (kilogram-force (kgf)) of at least 5 seconds each, with 30 seconds rest between them. The mean of the three trials will be used as the final strength value.

OTHER OUTCOMES:
Adverse events | immediately post-intervention
  Questionnaire for adverse events
Discomfort Rating (VAS) | immediately post-intervention
  The unpleasantness of the intervention will also be assessed using a 10 centimeters (cm) visual analogue scale (VAS), where 0 represents 'not unpleasant at all' and 10 represents 'the most unpleasant experience imaginable'.
Blinding Effectiveness Questionnaire | immediately post-intervention
  Blinding assessment for both the participant and the evaluator will be conducted at the end of each intervention. Blinding success will be evaluated using two consecutive questions, each offering five response options. The first question aims to discriminate between perceived percutaneous versus transcutaneous application, and the second question aims to distinguish between perceived active versus placebo stimulation.
  Participants and the evaluator will have no visual access to the device display during the intervention to maintain blinding

CONTACTS AND LOCATIONS:
Overall Officials: Diego Serrano Muñoz, Universidad de Castilla-La Man, Principal Investigator — Universidad de Castilla-La Mancha, Faculty of Physiotherapy and Nursing, Toledo, Spain
Locations (1):
- Universidad de Castilla La Mancha, Toledo, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No